CLINICAL TRIAL: NCT03611179
Title: Upfront Treatment With Chemotherapy and Bevacizumab in Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nada Hassan Salah (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Nada Hassan Salah, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bevacizumab in ovarian cancer
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Advanced Ovarian Cancer
Keywords: advanced ovarian cancer; upfront treatment; bevacizumab
MeSH Terms: interventions — Bevacizumab; Antineoplastic Agents

STUDY DESIGN:
Intervention Model Description: 40 patients diagnosed with advanced epithelial ovarian cancer presenting to Assiut university hospitals ,,the aim of the study is evaluation of response, survival and toxicity of upfront chemotherapy with Bevacizumab in those patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- advanced ovarian cancer cases (Experimental): patients with advanced ovarian cancer will receive Bevacizumab 15 mg/kg every 21 days with chemotherapy (Paclitaxel 175 mg/m2 & Carboplatin AUC 5 every 21 days)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — The chemotherapy regimen will be Paclitaxel (175 mg/m2 of body surface area) administered intravenously over 3 h, followed by carboplatin (area under the curve 5) over 1 h, with standard antiemetic and hypersensitivity medications.
  In patients who develop dose-limiting peripheral neuropathy or hypersensitivity, paclitaxel will be replaced with docetaxel (75 mg/m2), which is administered intravenously over 1 h.
  Bevacizumab (15 mg/kg bodyweight) administered intravenously initially over 90 min (if tolerated, this time can be reduced to 60 min, and could be further reduced to a minimum of 30 min)
  Other Names: Chemotherapy drugs

SUMMARY:
Our study aims at assessment of response, survival and toxicity of frontline treatment with chemotherapy and Bevacizumab in patients having advanced epithelial ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the most lethal gynecologic malignancy and is the fifth most common cause of cancer death in women .The majority of women with ovarian cancer are diagnosed with advanced-stage disease; only 15% of all cases are diagnosed with local disease. Risk factors for ovarian cancer include family history, nulliparity, lack of breast feeding, and infertility .

The GOG-0218 trial demonstrated that the use of bevacizumab in the front-line and maintenance setting improved progression free survival by 3.8 months when compared with conventional every-3-weeks carboplatin and paclitaxel.

The ICON-7 trial also aimed to compare the progression free survival and Overall survival in women who receive bevacizumab with carboplatin/paclitaxel and women receiving carboplatin/paclitaxel alone The final results of ICON7 were announced in 2013. Overall, the results showed no difference in overall survival between those in the group receiving bevacizumab han those in the group receiving no bevacizumab. However, for high-risk patients, who were most likely to have early disease progression, the results were positive and showed an improvement in overall survival of 4.8 months in the group who received bevacizumab.

Not only has the best route been intensely debated but the optimal timing of therapy has been and is currently being studied. Chemotherapy is usually given either only after primary debulking surgery or as both neoadjuvant chemotherapy before and after interval debulking surgery. recent trials have tried to determine which treatment timing is associated with better outcomes .

The aim of the study will be assessment of response, survival and toxicity of frontline treatment with chemotherapy and Bevacizumab in patients having advanced epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with advanced ovarian cancer by biopsy
* Age more than 18 years old
* Routine labs are within normal values ( CBC, renal function tests , liver function tests )
* Performance score 0-2
* FIGO stage II-IV
* Not having any contraindication to bevacizumab as : uncontrolled hypertension , bleeding tendency , ischaemic events
* Chemotherapy naïve.
* Informed consent

Exclusion Criteria:

* patients previously received chemotherapy or radiotherapy to any part of the abdomen or pelvis
* patients with uncontrolled infection
* patients with clinically significant cardiovascular disease
* patients with active bleeding or conditions associated with high risk of bleeding
* patients with history of CNS disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females diagnosed with ovarian cancer
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 years
  determination of time from starting treatment until first progression

CONTACTS AND LOCATIONS:
Overall Officials: mohammed A mekkawy, prof, Study Director — Assiut University; mohammed A hassan, lecturer, Study Director — Assiut University; hisham abo taleb, lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Aarnio M, Sankila R, Pukkala E, Salovaara R, Aaltonen LA, de la Chapelle A, Peltomaki P, Mecklin JP, Jarvinen HJ. Cancer risk in mutation carriers of DNA-mismatch-repair genes. Int J Cancer. 1999 Apr 12;81(2):214-8. doi: 10.1002/(sici)1097-0215(19990412)81:23.0.co;2-l. PMID 10188721
- [Background] Wright AA, Cronin A, Milne DE, Bookman MA, Burger RA, Cohn DE, Cristea MC, Griggs JJ, Keating NL, Levenback CF, Mantia-Smaldone G, Matulonis UA, Meyer LA, Niland JC, Weeks JC, O'Malley DM. Use and Effectiveness of Intraperitoneal Chemotherapy for Treatment of Ovarian Cancer. J Clin Oncol. 2015 Sep 10;33(26):2841-7. doi: 10.1200/JCO.2015.61.4776. Epub 2015 Aug 3. PMID 26240233